CLINICAL TRIAL: NCT01935336
Title: A Phase II Study of Ponatinib in Cohorts of Patients With Lung Cancer Preselected Using Different Candidate Predictive Biomarkers
Brief Title: Study of Ponatinib in Patients With Lung Cancer Preselected Using Different Candidate Predictive Biomarkers
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: Ariad Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 13-2002.cc; NCI-2013-01644 (Other: National Cancer Institute)
Record Dates: First submitted 2013-08-27; First posted 2013-09-05 (Estimated); Results first posted 2022-02-11 (Actual); Last update posted 2022-02-11 (Actual); Status verified 2022-01

CONDITIONS: Adenocarcinoma of the Lung; Extensive Stage Small Cell Lung Cancer; Limited Stage Small Cell Lung Cancer; Recurrent Non-small Cell Lung Cancer; Recurrent Small Cell Lung Cancer; Stage IIIA Non-small Cell Lung Cancer; Stage IIIB Non-small Cell Lung Cancer; Stage IV Non-small Cell Lung Cancer
Keywords: Lung Cancer; Malignancy; Predictive biomarkers
MeSH Terms: conditions — Adenocarcinoma of Lung; Carcinoma, Non-Small-Cell Lung; Small Cell Lung Carcinoma; Lung Neoplasms; Neoplasms | interventions — ponatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Ponatinib (Experimental): Patients receive ponatinib hydrochloride taken by mouth once or twice a day. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Ponatinib

INTERVENTIONS:
Drug: Ponatinib — Ponatinib 45mg taken by mouth each day at the same time with or without food
  Other Names: Iclusig; AP24534; Multitargeted tyrosine kinase inhibitor AP24534

SUMMARY:
This phase II trial studies how well ponatinib hydrochloride works in treating patients with stage III-IV lung cancer. Ponatinib hydrochloride may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth.

DETAILED DESCRIPTION:
This study will look at the safety and effectiveness of the investigational drug ponatinib in lung cancer. The investigators hope that ponatinib will work against tumors that have certain biomarkers. Therefore, the study will pre-screen patients for these certain biomarkers before enrolling them into the main treatment study. Different doses of ponatinib may be tested in this study.

ELIGIBILITY:
Inclusion Criteria:

* PART A: Patients must have histologically or cytologically confirmed locally advanced (after failure of local therapy) or metastatic lung cancer (any histology, except carcinoid) stage IIIa, IIIb or IV
* PART A: Existing formalin fixed paraffin embedded biopsy of the lung cancer with potentially sufficient material for analysis
* PART A: Non-small cell lung cancer (NSCLC) with adenocarcinoma histology must have been previously tested for both epidermal growth factor receptor (EGFR) mutations and anaplastic lymphoma kinase (ALK) rearrangements
* PART A: Able (physically and financially) to travel to University of Colorado for clinical trial treatment
* PART B: Patients must have histologically or cytologically confirmed locally advanced (after failure of local therapy) or metastatic lung cancer (any histology, except carcinoid) stage IIIa, IIIb or IV
* PART B: Patients must be proven to meet marker criteria (FGFR1 silver in situ hybridization (SISH) + in situ hybridization (ISH) +, FGFR1 SISH+ ISH negative [-ve], FGFR1 SISH-ve ISH+, FGFR1 SISH-ve ISH-ve [FGFR1 double negative cohort] or ret proto-oncogene [RET] FISH+) prior to enrollment into Part B (treatment); adenocarcinoma patients must be known to not possess either an EGFR mutation or an ALK rearrangement in their tumor (if positive for one, testing for both is not required)
* PART B: Patients must have measurable disease as per Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1
* PART B: Patients may have received any number of lines of prior therapy
* PART B: Life expectancy of >= 3 months
* PART B: Eastern Cooperative Oncology Group (ECOG) performance status =< 2 (Karnofsky >= 60%)
* PART B: Leukocytes >= 3,000/mcL
* PART B: Absolute neutrophil count >= 1,500/mcL
* PART B: Hemoglobin >= 9 g/dL
* PART B: Platelets >= 100,000/mcL
* PART B: Total bilirubin =< 1.5 x institutional upper limit of normal (ULN), unless due to Gilbert's syndrome
* PART B: Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 2.5 X ULN
* PART B: Creatinine =< 1.5 X ULN OR creatinine clearance >= 60 mL/min/1.73 m^2 for patients with creatinine levels above institutional normal
* PART B: Serum lipase =< 1.5 X ULN
* PART B: Serum amylase =< 1.5 X ULN
* PART B: Previous treatment related side-effects/adverse events must have resolved to at least grade 1 or, at the discretion of the investigator, select stable grade 2 toxicities (e.g. alopecia or fatigue) may be permissible if unchanging in grade for at least 3 months following discussion with the principal investigator (PI)
* PART B: Patients with central nervous system (CNS) metastases are eligible for enrollment if they have no overt evidence of neurological deficits, and are not requiring anti-epileptics or steroids to control their neurological symptoms; patients with known CNS metastases must have relevant CNS imaging performed approximately coincident with body imaging during response assessments
* PART B: The effects of ponatinib on the developing human fetus are unknown; for this reason women of child-bearing potential must have a negative urine or blood pregnancy test at screening for Part B; women of child-bearing potential and men must also have documented agreement to use adequate contraception (hormonal or barrier method of birth control; abstinence) from the time of screening until 30 days after the end of study treatment; should a woman become pregnant or suspect she is pregnant while she or her partner are participating in this study, they should inform the treating physician immediately
* PART B: Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* PART A: Known EGFR mutation and/or ALK rearrangement in NSCLC with adenocarcinoma histology
* PART B: No previous treatment with a standard or investigational anti-cancer agent within predicted 5 half-lives of the agent; or 28 days whichever is the shorter; if the plasma half-life is not known or the previous therapy was a monoclonal antibody then a 28 day washout period will be considered as the default requirement
* PART B: No previous or current exposure to other FGFR inhibitors in the FGFR-selected cohorts, or RET inhibitors in the RET selected cohorts
* PART B: Prior radiotherapy to proposed target lesions is not permitted unless completed more than 4 weeks prior to treatment within the study and that there has been documented progression at these sites; radiotherapy to non-target lesions is permitted within 2 weeks of study entry provided all acute effects of the radiotherapy have resolved to =< grade 1
* PART B: History of allergic or severe reactions attributed to compounds of similar chemical or biologic composition to ponatinib
* PART B: Ponatinib is a substrate for cytochrome P450, family 3, subfamily A, polypeptide 4/5 (CYP3A4/5), concurrent use with potent CYP3A4/5 inhibitors or inducers should be undertaken with caution
* PART B: History of clinically significant bleeding disorder
* PART B: History of acute pancreatitis within 1 year of study or history of chronic pancreatitis
* PART B: Uncontrolled hypertriglyceridemia (triglycerides > 450 mg/dL)
* PART B: Uncontrolled intercurrent illness including, but not limited to:

  * Ongoing or active infection requiring intravenous antibiotics
  * Psychiatric illness/social situations that would limit compliance with study requirements
  * Congestive heart failure, unstable angina pectoris, or myocardial infarction within the 3 months prior to enrollment in part B of the study
  * History of clinically significant (as determined by the treating medical doctor [MD]) cardiac arrhythmia (atrial or ventricular)
* PART B: Patients who have had major surgery within 28 days prior to entering the study or those who have not recovered from adverse events > grade 1 relating to the surgery
* PART B: Pregnant or breastfeeding women
* PART B: Patients with inability to take oral medications, or, in the investigator's opinion, gastrointestinal conditions or abnormalities likely to influence the absorption of oral medications
* PART B: Concomitant use of medications known to be associated with torsades-de-pointes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 171 (Actual)
Dates: Start 2013-09-24 (Actual); Primary Completion 2017-01 (Actual); Study Completion 2017-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ross D Camidge, MD, PhD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Cancer Center, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This is a biomarker driven clinical trial with prescreening for 4 molecular cohorts based on ISH and SISH positivity- FGFR1 ISH+/SISH+, FGFR1 ISH+/SISH-, FGFR1 ISH-/SISH+, and FGFR1 ISH-/SISH-; with the provision of testing for RET rearrangement in the double negative cohort.
  From Sep2013 to Nov2017, 171 patient samples were prescreened and resulted in 122 samples that had both SISH and ISH scores reportable. 4 of those patients signed main consent and were enrolled to treatment with ponatinib.
Pre-assignment Details: Tissue samples from patients were prescreened for markers. 171 samples were prescreened. Of these samples, biomarker results were obtained for 122 samples. Of the patients, from which these samples were derived, 4 patients were then enrolled on the study intervention, allocated to different arms based on their biomarker results. Unfortunately, due to poor tolerability and safety concerns regarding ponatinib after treating the first 4 patients, the trial stopped.
Groups:
- Ponatinib SISH+/ISH+: The pre-defined cutpoint for FGFR1 amplification (SISH+) was an average of at least four FGFR1 signals per nucleus (gene copy number) or FGFR1/CEP8 ratio ≥ 2.0.
  mRNA in situ hybridization (ISH) was performed on formalin-fixed paraffin embedded (FFPE) tumor tissue using the RNA scope 2.0 assay system. ISH scores were generated and recorded using the following scoring system at 200 × magnification: 0, no staining; 1, one to 3 dots per tumor cell; 2, 4 to 10 dots per tumor cell; 3, more than 10 dots per cell or presence of dot clusters in ≥1% and < 10% tumor cells; 4, ≥ 10% tumor cells with dot clusters as per the RNA scope system scoring guidelines.18 The pre-defined cutpoint for FGFR1 ISH positivity was a score of 3 or 4 per this scoring system.
- Ponatinib SISH+/ISH-: Please see details in Ponatinib SISH+/ISH+ for the definition of SISH positivity and ISH positivity.
  Subjects in this group are those with SISH positive and ISH negative.
- Ponatinib SISH-/ISH+: Please see details in Ponatinib SISH+/ISH+ for the definition of SISH positivity and ISH positivity.
  Subjects in this group with a negative SISH and a positive ISH
- Ponatinib SISH-/ISH-: Please see details in Ponatinib SISH+/ISH+ for the definition of SISH positivity and ISH positivity.
  Subjects in this group with a negative SISH and a negative ISH
Period: Overall Study
Arm/Group | Ponatinib SISH+/ISH+ | Ponatinib SISH+/ISH- | Ponatinib SISH-/ISH+ | Ponatinib SISH-/ISH-
Started | 6 (Only one subject was treated due to the black box warning RE: ponatinib-associated vascular issues. The protocol was modified with additional inclusion and exclusion criteria, which severely limited the number of cases treated with the drug) | 3 (no subjects were treated in this arm) | 47 (Only three subjects were treated due to the black box warning RE: ponatinib-associated vascular issues. The protocol was modified with additional inclusion and exclusion criteria, which severely limited the number of cases treated with the drug) | 66 (No subjects were treated in this arm)
Started Treatment | 1 | 0 | 3 | 0
Completed | 0 | 0 | 0 | 0
Not Completed | 6 | 3 | 47 | 66
Not completed — Adverse Event | 1 | 0 | 0 | 0
Not completed — Progressive disease | 5 | 3 | 47 | 66

BASELINE CHARACTERISTICS:
Population: 171 subjects were pre-screen consented to request and submit tissue for ISH and SISH scoring. 122 of 171 subjects received ISH/SISH results and of those 122 subjects who received ISH/SISH results, 4 were main consented and enrolled to actual treatment with ponatinib.
Groups:
- Total: Total of all reporting groups
Arm/Group | Ponatinib SISH+/ISH+ | Ponatinib SISH+/ISH- | Ponatinib SISH-/ISH+ | Ponatinib SISH-/ISH- | Total
Number analyzed (Participants) | 6 | 3 | 47 | 66 | 122
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 66.9 [64.88 to 72.38] | 68.80 [67.05 to 69.15] | 65.70 [57.50 to 72.55] | 63.50 [58.05 to 70.70] | 65.0 [58.05 to 72.45]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 26 | 33 | 61
  Male | 5 | 2 | 21 | 33 | 61
Smoking PY [Median (Inter-Quartile Range); unit: Pack/year] | 37.5 [31.35 to 51.25] | 57 [45 to 68.5] | 30 [17.5 to 50.0] | 30 [9 to 42.94] | 30.73 [11.3 to 45]
Sites of metastases (soft tissue) [Count of Participants; unit: Participants]
  Yes | 0 | 0 | 6 | 4 | 10
  No | 6 | 3 | 41 | 62 | 112
Histology [Count of Participants; unit: Participants]
  Adenoca | 2 | 2 | 28 | 48 | 80
  Squamous | 1 | 1 | 11 | 8 | 21
  Small cell | 3 | 0 | 8 | 10 | 21
KRAS [Count of Participants; unit: Participants]
  No | 3 | 3 | 22 | 26 | 54
  Yes | 0 | 0 | 16 | 28 | 44
  unevaluable | 3 | 0 | 9 | 12 | 24

OUTCOME MEASURES:

1. Primary Outcome: Biomarker FGFR1 (ISH/SISH) Score (Part A)
Description: Biomarker prevalence and its 95% (exact) confidence interval (CI) among the screening patients and for different histologies will be reported. Molecular cohorts for ISH and SISH positivity: FGFR1 ISH+/SISH+, FGFR1 ISH+/SISH-, FGFR1 ISH-/SISH+, and FGFR1 ISH-/SISH-
Time Frame: Baseline
Population: 171 cases were prescreened. Among them, 122 cases had both SISH and ISH scores reported, one case had only SISH and four cases had only ISH reported, and 44 cases lacked both SISH and ISH scores, resulting in 123 cases with SISH and 126 cases with ISH. Please note that the 126 cases with ISH scores were displayed in two different ways, one was based on ISH<1% vs >+1% (columns 3 and 4 above), and the other was based on ISH<20% vs >=20% (columns 5 and 6).
Measure: Mean (95% Confidence Interval); unit: gene copy number
Groups:
- SISH-: Less than four FGFR1 signals per nucleus (gene copy number) or FGFR1/CEP8 ratio ≥ 2.0
- SISH+: At least four FGFR1 signals per nucleus (gene copy number) or FGFR1/CEP8 ratio ≥ 2.0
- ISH-(<1%): mRNA in situ hybridization with dot clusters per tumor <1%
- ISH+(>=1%): mRNA in situ hybridization with dot clusters 1%=<per tumor <10%
- ISH<20%: mRNA in situ hybridization with dot clusters 10%=<per tumor <20%
- ISH>=20%: mRNA in situ hybridization with dot clusters 1per tumor >=20%
Arm/Group | SISH- | SISH+ | ISH-(<1%) | ISH+(>=1%) | ISH<20% | ISH>=20%
Number analyzed (Participants) | 114 | 9 | 73 | 53 | 97 | 29
gene copy number | 0.93 [0.87 to 0.97] | 0.07 [0.03 to 0.134] | 0.579 [0.488 to 0.667] | 0.42 [0.333 to 0.512] | 0.77 [0.686 to 0.84] | 0.23 [0.16 to 0.31]

2. Primary Outcome: Overlapping Frequency of FGFR1 (ISH/SISH) Biomarkers (Part A)
Description: Overlapping frequency and its 95% CI between biomarkers among the screening patients and for different histologies will also be reported.
Time Frame: Baseline
Population: 171 subjects were pre-screen consented to request and submit tissue for ISH and SISH scoring. 122 of 171 subjects received ISH/SISH results and of those 122 subjects who received ISH/SISH results, 4 were enrolled to actual treatment with ponatinib. The number reported here are the eligible number of subjects in each pre-defined category.
Measure: Mean (95% Confidence Interval); unit: gene copy number
Arm/Group | Ponatinib SISH+/ISH+ | Ponatinib SISH+/ISH- | Ponatinib SISH-/ISH+ | Ponatinib SISH-/ISH-
Number analyzed (Participants) | 6 | 3 | 47 | 66
gene copy number | 0.049 [0.018 to 0.104] | 0.0246 [0.005 to 0.070] | 0.385 [0.299 to 0.478] | 0.541 [0.448 to 0.632]

3. Primary Outcome: Objective Response Rate (ORR) Per RECIST v1.1 (Part B)
Description: Evaluated using Fisher's exact test with a descriptive p-value. Summarized using binomial proportions with 95% exact binomial confidence intervals.
Time Frame: From date of first dose until date of Disease Progression or death (up to 153 days), whichever occurred first
Population: A total of 4 subjects were treated, where the 3 SISH-/ISH+ all with RET-, due to the safety concern of ponatinib and the change of inclusion and exclusion criteria.
Measure: Count of Participants; unit: Participants
Arm/Group | Ponatinib SISH+/ISH+ | Ponatinib SISH+/ISH- | Ponatinib SISH-/ISH+ | Ponatinib SISH-/ISH-
Number analyzed (Participants) | 1 | 0 | 3 | 0
Participants | 0 | 0 | 0 | 0

4. Secondary Outcome: Incidence of Adverse Events, Graded According to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) v4.0
Description: Adverse events will be tabulated per participant, per organ, and per visit.
Time Frame: From date of first dose until date of Disease Progression (up to 153 days). Assessed at Day 1, Day 8, Day 15 of each 28 day cycle)
Population: Due to the safety warning of Ponatinib and the adjusted inclusion and exclusion criteria, the study only treated 4 subjects in total.
Measure: Number; unit: participants
Arm/Group | Ponatinib SISH+/ISH+ | Ponatinib SISH+/ISH- | Ponatinib SISH-/ISH+ | Ponatinib SISH-/ISH-
Number analyzed (Participants) | 1 | 0 | 3 | 0
participants
  Grade 3 | 0 |  | 2 |
  Gr 3 fibrillation or febrile neutropenia or platelets | 1 |  | 2 |

ADVERSE EVENTS:
Time Frame: During the first year post treatment
Description: The number at risk for all-cause mortality is 4 The number at risk for SAE was 4. There were 75% SAEs.
Arm/Group | Ponatinib SISH+/ISH+ | Ponatinib SISH+/ISH- | Ponatinib SISH-/ISH+ | Ponatinib SISH-/ISH-
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/0 | 0/3 | 0/0
Serious Adverse Events (participants affected / at risk) | 1/1 | 0/0 | 2/3 | 0/0
Other Adverse Events (participants affected / at risk) | 1/1 | 0/0 | 2/3 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ponatinib SISH+/ISH+ (N=1) | Ponatinib SISH+/ISH- (N=0) | Ponatinib SISH-/ISH+ (N=3) | Ponatinib SISH-/ISH- (N=0)
Grade 3 AE (Gastrointestinal disorders) | 1 (1) | NA | 2 (2) | NA — Febrile neutropenia, Bowel perforation, Hyponatremia
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ponatinib SISH+/ISH+ (N=1) | Ponatinib SISH+/ISH- (N=0) | Ponatinib SISH-/ISH+ (N=3) | Ponatinib SISH-/ISH- (N=0)
Grade 2 hypertension (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 2 (3) | 0 (0)
Grade 2 thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
Due to poor tolerability and safety concerns regarding ponatinib after treating the first few patients, the study did not reach its accrual target (N~70) for the treatment portion of this study and could not confirm or refute the null hypothesis (needed a minimum of 12 patients treated). This study prescreened a more heterogeneous population. As a result, all four patients that were enrolled onto the ponatinib treatment arm had either squamous or poorly differentiated lung cancer.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2017-08-02): https://cdn.clinicaltrials.gov/large-docs/36/NCT01935336/Prot_SAP_ICF_000.pdf